CLINICAL TRIAL: NCT01541228
Title: Clinical Effect of Photodynamic Treatment When Treating Actinic Keratoses With Different Light Doses
Brief Title: Photodynamic Treatment of Actinic Keratoses With Different Light Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Evelina Buinauskaite, Principal investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BE-2-60
Record Dates: First submitted 2012-02-14; First posted 2012-02-29 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; photodynamic therapy; 5-aminolevulinic acid
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Active Comparator): Patients with actinic keratosis (AK) on the left and right sides of face/scalp region treated with photodynamic therapy using 20% 5-aminolevulinic acid.
  Interventions: Device: Photodynamic therapy with light dose of 70 J/cm2 using a broad-band red light source
- Group II (Active Comparator): Patients with actinic keratosis (AK) on the left and right sides of the face/scalp region treated with photodynamic therapy using 20% 5-aminolevulinic acid.
  Interventions: Procedure: Photodynamic therapy with 100J/cm2 light dose using a broad-band red light source

INTERVENTIONS:
Device: Photodynamic therapy with light dose of 70 J/cm2 using a broad-band red light source — Patients take part in intraindividual (left-right) comparison study when having at least 2 non-hyperkeratotic actinic keratoses (AK) on the left and right sides of the face/scalp.
  Punch biopsies in 3.5 millimetres diameter performed to confirm the diagnosis of AK.
  Patients randomized so that half of them would receive a light dose of 70J/cm2 as their first split face/scalp treatment on the left side. Photodynamic therapy with the light dose of 70 J/cm2 using a broad-band red light source (570-670 nm,Curelight®, PhotoCure, Oslo, Norway) and 20% 5-ALA. Treatment repeated twice with two weeks interval.
  Arms: Group I
Procedure: Photodynamic therapy with 100J/cm2 light dose using a broad-band red light source — Patients take part in intraindividual (left-right) comparison study when having at least 2 non-hyperkeratotic actinic keratoses (AK) on the left and right sides of the face/scalp. Punch biopsies in 3.5 millimetres diameter performed to confirm the diagnosis of AK.
  Patients randomized so that half of them would receive a light dose of 100J/cm2 as their first split face/scalp treatment on the left side. Photodynamic therapy with the light dose of 70 J/cm2 using a broad-band red light source (570-670 nm,Curelight®, PhotoCure, Oslo, Norway) and 20% 5-ALA.Treatment repeated twice with two weeks interval.
  Arms: Group II

SUMMARY:
Aim of the study: To evaluate clinical effectiveness of two different light doses when treating actinic keratoses with photodynamic therapy with 20% 5-aminolevulinic acid.

DETAILED DESCRIPTION:
To determine and compare clinical and histological effectiveness of different (70 J/cm2 ir 100 J/cm2) light doses when treating actinic keratoses with photodynamic therapy.

To determine pain intensity during photodynamic therapy with visual analogue scale and factors influencing pain during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject older than 50 years.
2. Subject has to read Patient Information Sheet and read and sign the Informed Consent form prior to any study related procedure.
3. AK with the largest diameter ≤3 cm (measuring the longest axis).
4. 2 or more AK with symmetrical distribution on the face or scalp.
5. Clinically and histologically confirmed AK of grade I or II.
6. Subject must be willing and capable of cooperating to the extent and degree required by the protocol.
7. Patient is not the subject of the administrative or legal judicial proceeding.
8. Subject has social health security required by laws of health care institutions.

Exclusion Criteria:

1. Patients with more than 5 AK in the planned treatment area.
2. A recurrent AK: AK that has been previously treated in the study area.
3. Very hyperkeratotic, grade 3 (on a 0-3 scale) AK lesions among the target lesions.
4. AK located on the nose.
5. Other skin lesions (diseases) in the tumor study area.
6. Subject with known hereditary basal cell carcinoma syndromes (Gorlin-Goltz, Basex-Dupre-Christol et al.).
7. Subject with a history of cutaneous photosensitization or porphyria or Xeroderma pigmentosum, hypersensitivity to porphyrins, or photodermatosis.
8. Subject who had received photosensitizing drugs 30 days before study start.
9. Subjects who had received immunomodulatory or immunosuppressive therapies, including systemic and topical steroids, imiquimod or solaraze, interferon and acitretin 6 months prior to study treatment initiation.
10. Subject who had participated in another investigational drug or device research study within 30 days of enrolment.
11. Subject had received in the study area laser resurfacing, chemical peels, topical application fluorouracil or other drugs for the treatment of AKs within 2 months before study entry.
12. Subject with known hypersensitivity to 5-aminolevulinc acid, a similar compound or excipients of the cream.
13. Subject with known status after organ transplantation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Clinically cleared actinic keratosis with histological evaluation when clinically suspicious for relapse | 3 months
  All treated actinic keratoses evaluated by two investigators for clinical/histological relapse at months 1, 3, 6, 12, 24 after treatment

SECONDARY OUTCOMES:
Pain during the treatment | 2 years
  Patients inform a present investigator about pain severity at the beginning, in the middle, at the end of the session and move a counter of visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Evelina Buinauskaite, MD, Principal Investigator — Lithuanian University of Health Sciences, Medical Academy, Department of Skin and Venereal Diseases; Skaidra Valiukeviciene, Prof., Study Chair — 1Lithuanian University of Health Sciences, Medical Academy, Department of Skin and Venereal Diseases
Locations (1):
- Department of Skin and Venereal Diseases, Lithuanian University of Health Sciences, Medical Academy, Kaunas, Eiveniu Saint 2, Lithuania

REFERENCES:
- [Result] Buinauskaite E, Zalinkevicius R, Buinauskiene J, Valiukeviciene S. Pain during topical photodynamic therapy of actinic keratoses with 5-aminolevulinic acid and red light source: randomized controlled trial. Photodermatol Photoimmunol Photomed. 2013 Aug;29(4):173-81. doi: 10.1111/phpp.12044. PMID 23815349